CLINICAL TRIAL: NCT06299904
Title: Effect of Modified Air-pulse Stimulation on Tracheotomised Patients With Dysphagia After Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: stroke
Record Dates: First submitted 2024-03-01; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Sham Comparator): Based on receiving personalized swallowing rehabilitation training, the control group received traditional air-pulse stimulation therapy.
  Interventions: Behavioral: Conventional air-pulse stimulation
- trial group (Experimental): The trial group received modified air-pulse stimulation therapy mediated by flexible endoscopy.
  Interventions: Behavioral: Modified Air-pulse Stimulation

INTERVENTIONS:
Behavioral: Modified Air-pulse Stimulation — Connected the oxygen humidification bottle to a fibreoptic endoscope, then inserted the terminal into the nasal cavity and the pulse sensation stimulation generated by oxygen was transmitted through the internal port of the fibreoptic endoscope to the anterior wall of the pyriform recess or to the folds of the arytenoepiglottis. (5 min once a day for 2 weeks)
  Arms: trial group
Behavioral: Conventional air-pulse stimulation — The terminal airway of the air pulse was placed in the oral cavity, specifically in the patient's palatoglossal arch, pharyngeal posterior wall, tongue base, and other areas. The airbag was quickly squeezed to generate airflow and stimulate the mucosa.(5 min once a day for 2 weeks)
  Arms: control group

SUMMARY:
To evaluate the efficacy of flexible endoscopy-mediated modified air-pulse stimulation in restoring of swallowing function in this group of patients.Forty-two subacute stroke patients with tracheotomy and dysphagia need to be recruited and divided into a control group of 21 cases and a trial group of 21 cases. On the basis of receiving personalized swallowing rehabilitation training, the control group received traditional air-pulse stimulation therapy, while the trial group received modified air-pulse stimulation therapy mediated by flexible endoscopy. Murray secretion scale (MSS), penetration-aspiration scale (PAS) and spontaneous swallowing frequency were used to assess dysphagia. Moreover, clinical pulmonary infection score (CPIS) was used for evaluating the degree of pneumonia, hemoglobin(Hb) and serum prealbumin (PAB) were used to assess the nutritional status of patients.

ELIGIBILITY:
Inclusion Criteria:

* patients who met the diagnostic criteria for stroke formulated in the 4th National Academic Conference on Cerebrovascular disease;
* patients with relatively stable vital signs, with a NIHSS score of 21 points;
* patients with tracheotomy accompanied by dysphagia;
* no previous history of dysphagia;
* age ≥ 30 years and ≤80 years;
* informed consent signed by the patient and his family.

Exclusion Criteria:

* patients with medullary haemorrhage/infarction;
* patients that experienced cerebral hernia and recurrent stroke;
* patients with unstable arrhythmia, fever, infection, severe restlessness and inability to cooperate with treatment;
* patients with gastro-oesophageal reflux, bilateral paralysis of the vocal cord, laryngopharyngeal stenosis/haemorrhage/tumour;
* patients in which there was an inability to accurately locate epiglottis and arytenoid cartilage due to throat disease;
* patients with a history of epilepsy or risk of seizures.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
the score of Fiberoptic endoscopic examination of swallowing (FEES) | 2 weeks
  Fiberoptic endoscopic examination of swallowing
the score of Murray's secretion scale (MSS) | 2 weeks
  MSS
the score of penetration-aspiration scale (PAS) | 2 weeks
  PAS

SECONDARY OUTCOMES:
the score of Clinical Pulmonary Infection Score (CPIS) | 2 weeks
  CPIS

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital of Dalian Medical University, Dalian, Liaoning, China